CLINICAL TRIAL: NCT00514215
Title: Percutaneous Cryotherapy and Aerosolized GM-CSF for Pulmonary Metastases and Primary Lung Cancer
Brief Title: Cryotherapy and GM-CSF in Treating Patients With Lung Metastases or Primary Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Littrup, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000559667; P30CA022453 (NIH); WSU-C-2795; WSU-HIC-050304M1(R)F
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Kidney Cancer; Lung Cancer; Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: lung metastases; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; recurrent renal cell cancer; stage IV renal cell cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Kidney Neoplasms; Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; Flow Cytometry; Immunoenzyme Techniques; Biopsy; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sargramostim, Flow Cytometry, Biopsy. Cryosurgery (Experimental): Sargramostim-250 μg, inhaled, two times a day, on days 4-10 and days 36-42 Flow cytometry-Days 1 & 32 Immunoenzyme technique-Days 1 & 32 CT guided biopsy-Days 1 & 32 Cryosurgery-Days 1 and 32
  Interventions: Biological: sargramostim; Other: flow cytometry; Other: immunoenzyme technique; Procedure: biopsy; Procedure: cryosurgery

INTERVENTIONS:
Biological: sargramostim — 250 μg, inhaled, two times a day, on days 4-10 and days 36-42
  Other Names: GM-CSF (Granulocyte-Macrophage Colony Stimulating Factor); Leukine
Other: flow cytometry — Days 1 & 32
Other: immunoenzyme technique — Days 1 & 32
Procedure: biopsy — CT guided biopsy on days 1 & 32
Procedure: cryosurgery — Days 1 and 32

SUMMARY:
RATIONALE: Cryotherapy kills tumor cells by freezing them. Giving an injection of GM-CSF before cryotherapy and inhaling GM-CSF after cryotherapy may interfere with the growth of tumor cells and shrink the tumor. Giving cryotherapy together with GM-CSF may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cryotherapy together with GM-CSF works in treating patients with lung metastases or primary lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether percutaneous cryotherapy in combination with aerosolized sargramostim (GM-CSF) has any demonstrable immunologic effect in patients with pulmonary metastases or primary lung cancer.
* Determine whether any systemic immune response is detectable by the combination of cryotherapy as the antigen presentation source and GM-CSF as the immunologic adjuvant.
* Determine whether low morbidities will be maintained in patients treated with this regimen.
* Determine whether effective immunization is associated with a drop in CD4+, CD25+, LTP(TGF-β1)+, Tr cells as measured by flow cytometry or ELISPOT assay for TGF-β1-secreting cells.

Secondary

* Determine clinical response (i.e., tumor control in the dominant masses undergoing cryotherapy or in other metastatic sites) as measured by CT criteria.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients undergo CT-guided core biopsy of a dominant lung mass and placement of at least 2 cryoprobes. Prior to initiating the freeze, patients receive an interstitial injection of sargramostim (GM-CSF) near the tumor. Patients then undergo percutaneous cryotherapy over 2 hours utilizing a freeze-thaw-freeze cycle. Beginning within 3 days of cryotherapy, patients receive aerosolized GM-CSF twice daily for 1 week. Beginning on day 32, patients may elect to undergo a second course of treatment as described above in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and tumor tissue collection at baseline and periodically during study for immunological correlative studies. Peripheral blood mononuclear cells isolated from blood samples are analyzed for antigen-specific CD4-positive or CD8-positive T-cell response by flow cytometry or by TGF-β1 ELISPOT assay to measure TGF-β1- secreting cells. Tumor cell lysates extracted from tumor samples are pulsed with autologous dendritic cells and analyzed by ELISPOT assay to measure T-cell reactivity in tumor specimens.

After completion of study therapy, patients are followed at 6 and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Primary non-small cell lung cancer (NSCLC)

    * Any stage nonoperative NSCLC or patient refuses surgery
  * Any cancer with pulmonary metastatic disease (including renal cell cancer)

    * Stage IV disease (any T, any N, M1)
* Must have 1-10 pulmonary or mediastinal masses meeting the following criteria:

  * At least 1 mass is appropriate for 2 sessions of core biopsy and cryotherapy with relatively easy access/low risk in nonoperative patients (or those refusing surgery)
  * The two dominant masses are defined as either the largest and/or those that may cause imminent morbidity from continued local progression, thereby potentially benefiting from thoracic cryotherapy alone
  * Optimal tumor size > 1.0 cm

    * Dominant masses up to 6 cm in diameter may be considered if thorough cryotherapy coverage can be anticipated with minimal additional treatment morbidity
* Measurable disease, defined as tridimensional measurements of up to 6 different pulmonary or mediastinal masses ≥ 0.5 cm by CT scan
* No active pleural effusion that could be related to respiratory infection or requires further work-up
* No untreated and/or unstable brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 12 weeks
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 50,000/mm³
* INR < 1.5 (i.e., normal PT/PTT)
* Hemoglobin ≥ 8.0 g/dL
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Satisfactory pulmonary function test as determined by supervising oncologist, thoracic surgeon, or pulmonologist
* Not pregnant or lactating
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Inactive history of cancer allowed if the patient has been disease-free for > 2 years
* No serious medical or psychiatric illnesses that would preclude informed consent or limit survival to < 12 wks
* No uncontrollable cough or inability to lie flat
* No New York Heart Association class III or IV heart disease
* No known immunodeficiency state
* No uncontrolled infection
* No uncontrolled coagulopathy or bleeding diathesis
* No advance directive that would prevent the investigator from treating the participant in the event of a complication occurring during or after the procedure
* No medical contraindication or potential problem that would preclude protocol compliance

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 4 weeks since prior radiotherapy
* More than 2 weeks since prior corticosteroids
* More than 1 week since prior parenteral antibiotics
* At least 1 week since prior aspirin or aspirin-like medications
* At least 3 days since prior warfarin, clopidogrel bisulfate, or similar compounds
* No concurrent GM-CSF other than study drug
* No concurrent G-CSF
* No concurrent radiotherapy
* No concurrent glucocorticosteroids
* No concurrent parenteral antibiotics
* No concurrent immunosuppressive agents
* No concurrent drugs that cause bleeding tendencies
* No other concurrent biologic therapy, immunotherapy, radiotherapy, or chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Littrup, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sargramostim, Flow Cytometry, Biopsy. Cryosurgery
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sargramostim, Flow Cytometry, Biopsy. Cryosurgery
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 55 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Response as Measured by ELISPOT Assay and Flow Cytometry
Description: CT-guided biopsy & Peritumoral GM-CSF. a CR was defined as involution of the prior tumor and/or ablation site to only a thin, non-enhancing scar within the pulmonary parenchyma on enhanced chest CT. A PR was defined as incomplete resolution of an otherwise thoroughly hypovascular resolving ablation zone which had reached a diameter smaller than the original tumor size. Stable disease (SD) reflects no significant change in size of ablation site and/or overall tumor burden, while the standard definition for progressive disease (PD) remains as evidence of neTw or growing tumors.
Time Frame: Days 1 & 32
Population: Patients who had metastatic Renal Cell carcinoma
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim, Flow Cytometry, Biopsy. Cryosurgery
Number analyzed (Participants) | 6
Participants
  Complete Response | 1
  Partial Response | 3
  Progressive Disease | 2

2. Secondary Outcome: Clinical Response as Measured by CT Criteria
Description: CT-guided biopsy. a CR was defined as involution of the prior tumor and/or ablation site to only a thin, non-enhancing scar within the pulmonary parenchyma on enhanced chest CT. A PR was defined as incomplete resolution of an otherwise thoroughly hypovascular resolving ablation zone which had reached a diameter smaller than the original tumor size. Stable disease (SD) reflects no significant change in size of ablation site and/or overall tumor burden, while the standard definition for progressive disease (PD) remains as evidence of neTw or growing tumors.
Time Frame: Days 1 & 32
Population: only those with metastatic Renal Cell carcinoma
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim, Flow Cytometry, Biopsy. Cryosurgery
Number analyzed (Participants) | 6
Participants
  Complete Response | 1
  Partial Response | 3
  Progressive Disease | 2

3. Secondary Outcome: Toxicity of Grade 1 or Higher
Description: Number of Participants with Toxicity of Grade 1 or Higher as defined by CTCAE v2
Time Frame: Days 11, 32, 43, & 63
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim, Flow Cytometry, Biopsy. Cryosurgery
Number analyzed (Participants) | 8
Participants
  Alergic Reaction | 1
  Allergic rhinitis | 2
  Anemia | 1
  Anorexia | 1
  Atelectasis | 1
  Bronchospasm, wheezing | 1
  Chest Pain (noncardiac, nonpleuritic) | 1
  Chest wall pain | 6
  Cough | 7
  Decreased platelets | 1
  Dizziness | 1
  Dyspnea | 4
  Fatigue | 4
  Hemoptysis | 1
  Hemorrhage, pulmonary lung (hemoptysis) | 4
  Hyperglycemia | 1
  Low grade fever | 1
  Lymphopenia | 2
  Nausea | 1
  Pain at incision site | 1
  Pain-upper resp. throat | 2
  Platelets Low | 1
  Pneumothorax | 4
  Sensory Neuropathy | 1
  Shortness of Breath | 1
  Sweating | 1
  Thrombocytopenia | 1
  Vomiting | 1

4. Secondary Outcome: Immune Function and Cancer-specific Response
Description: Number of Participants with CT-guided biopsy & Peritumoral GM-CSF. The number of IFNγ secreting T-cells was measured by a direct EliSpots at 10:1 E:T ratio to define the kinetics of the CTL responses from pre-CI to day 63 post CI.
Time Frame: Days 1 & 63
Population: only those with metastatic Renal Cell carcinoma
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim, Flow Cytometry, Biopsy. Cryosurgery
Number analyzed (Participants) | 6
Participants
  increase of IFN gamma secreting T cells | 4
  elevated antibody levels | 4
  Increased anti-RC-2+KCI-18 serum antibodies | 4

ADVERSE EVENTS:
Arm/Group | Sargramostim, Flow Cytometry, Biopsy. Cryosurgery
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sargramostim, Flow Cytometry, Biopsy. Cryosurgery (N=8)
Allergic Reaction (Immune system disorders) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Pain (noncardiac, nonpleuritic) (General disorders) | 1 (1)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 6 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Decreased Platelets ( thrombocytopenia) (Blood and lymphatic system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Fatigue (General disorders) | 4 (4)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage, pulmonary lung (hemoptysis) (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Low grade fever (General disorders) | 1 (1)
Lymphopenia (low lever of lymphocytes) (Investigations) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain at incision site (General disorders) | 1 (1)
Pain - Upper Respiratory throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Platelets (low count, thrombocytopenia) (Investigations) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Sensory Neuropathy (Nervous system disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No